CLINICAL TRIAL: NCT05049148
Title: Observation of Platelets in Primary and Secondary Tumors of the Central Nervous System and Association With Survival: a Prospective Cohort Study
Brief Title: Platelets Activation in Brain Neoplasms
Acronym: Platon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBN_2021_6
Record Dates: First submitted 2021-08-18; First posted 2021-09-17 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Glioma; Blood Platelets; Inflammation; Brain Neoplasms
Keywords: Platelets activation
MeSH Terms: conditions — Glioma; Inflammation; Brain Neoplasms | interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients requirering brain/medullary tumors excision (Other): All patients requirering a surgery for brain or medullar excision
  Interventions: Other: Platelet count in excised tumors

INTERVENTIONS:
Other: Platelet count in excised tumors — Tumors excised in patients requirering a brain or medullary surgery will be assess to determine their platelet count.

SUMMARY:
Platelets are primarily known for their central role in primary hemostasis. However, they are increasingly recognized for their participation in various non-hemostatic processes, such as cancer progression and clinical expression. Experimental and clinical data indicate that the involvement of platelets in the pathophysiology of cancer goes far beyond the realm of cancer-associated thrombosis.

Several experimental studies have shown that platelets can promote the metastatic process by various mechanisms. However, while it has been shown in vitro that direct contact with platelets initiates tumor cells for metastasis, it remains unclear whether such contacts occur in solid tumors. In addition to their ability to promote metastasis, platelets have been shown to stimulate angiogenesis and play a crucial role in lymphangiogenesis.

Considering that blood vessels, lymphatics and immune cells are major components of the tumor ecosystem, our hypothesis is that platelets contribute to the development and / or regulation of the tumor microenvironment. This is because platelets stabilize tumor blood vessels by permanently repairing vascular damage caused by immune cells infiltrating tumors. Targeting platelets destabilizes tumor vessels, causing intra-tumor hemorrhage, which allows intra-tumor accumulation of intravenously administered anti-tumor drugs such as paclitaxel and improves their efficacy.

Studies have also reported the role of platelets in several pathogenic mechanisms of cancer: thrombocytosis is a paraneoplastic syndrome which suggests a poor prognosis in patients with solid tumors; a negative correlation between the platelet count and the response to chemotherapy has been reported in several types of cancer; histological analyzes of esophageal cancer suggested a possible association between the presence of platelets in the tumor stroma and the level of tumor lymphangiogenesis and lymphovascular invasion; finally, a recent study reported the expression of one of the main targets of immunotherapies, PD-L1, on the platelets of patients suffering from different types of solid cancers.

All of these data support our hypothesis that platelets are components and / or regulators of the tumor microenvironment and therefore potential targets for the improvement of anti-tumor therapies. In this context, the objectives of our project are to determine whether platelets are components of the microenvironment of tumors of the central nervous system, and to study the possible correlations between the intratumoral presence of platelets and the evolution of patients with central nervous system tumors

DETAILED DESCRIPTION:
This is a descriptive study that did not include any intervention other than tumor tissue preservation and blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Patient to undergo excision or biopsy of a brain or medullary tumor
* Patient over 18 years old
* Express consent to participate in the study
* Affiliate member of the Social Security system

Exclusion Criteria:

* Tumor sample volume not allowing the performance of additional analyzes
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Platelet detection in excised brain/medurally tumors | 1 hour
  biopsy: Presence of neo-vessels

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOURDILLON, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A De Rothschild, Paris, France